CLINICAL TRIAL: NCT01274351
Title: A Phase II Multi-center, Open-label, Non-randomized Study of Nilotinib as First Line Treatment in Adult Patients With Newly Diagnosed Philadelphia Chromosome Positive (Ph+) Chronic Myelogenous Leukemia in Chronic Phase (CML-CP)
Brief Title: Study of Nilotinib as First Line Treatment in Philadelphia Chromosome Positive(Ph+) Chronic Myelogenous Leukemia in Chronic Phase (CML-CP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107ETR02
Record Dates: First submitted 2011-01-04; First posted 2011-01-11 (Estimated); Results first posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: First line treatment; newly diagnosed; Philadelphia chromosome positive; Chronic Myelogenous Leukemia; Ph+; CML-CP; major molecular response; Social risk
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nilotinib (Experimental): administered orally at a dose of 300 mg twice daily for 24 months
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — administered orally at a dose of 300 mg twice daily for 24 months
  Other Names: Tasigna, AMN107

SUMMARY:
The study was a local multicentric, open-label, non-randomized phase II study of nilotinib as a first line treatment in adult patients with newly-diagnosed Philadelphia chromosome-positive (Ph+) and chronic phase myeloid leukemia (CML-CP).

DETAILED DESCRIPTION:
This was a multicenter, open-label, single-arm, phase 2 study of nilotinib as a frontline treatment for patients with Ph+ CMLCP. All patients received oral nilotinib 300 mg twice daily for a planned treatment duration of 24 months or until early discontinuation.

The primary efficacy end point was the cumulative rate of Major Molecular Response (MMR) in all participants by 12 months. Secondary efficacy end points included the rate of Complete Cytogenic Response (CCyR) at 6 and 12 months; cumulative rates of MMR up to 24 months; time to and durability of MMR; and cumulative rate of Complete Haematologic Response (CHR) by 12 months.

Patient evaluations, including hematologic assessments, were conducted every 15 days during the first 3 months, monthly until month 12, and then every 3 months until the end of the study (24 months). All efficacy analyses were performed in the intent-to treat population.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* First cytogenetic diagnosis of CML-CP with cytogenetic confirmation of Philadelphia chromosome of (9;22) translocations within 6 months. Standard conventional cytogenetic analysis must be performed.
* Previously untreated for CML, except for hydroxyurea and/or anagrelide (except imatinib treatment for max. 31 days long)
* Adequate end organ function with following laboratory criteria: total bilirubin < 1.5 x upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x upper limit of normal (ULN); creatinine < 1.5 x upper limit of normal (ULN); serum amylase and lipase ≤ 1.5 x upper limit of normal (ULN); alkaline phosphatase ≤ 2.5 x upper limit of normal (ULN) unless considered tumor related
* Serum potassium, magnesium, and phosphorus levels are equal or above the lower limit of normal prior to the first dose of study medication

Exclusion Criteria:

* Treatment with tyrosine kinase inhibitor(s) prior to study (in emergent cases where the patient requires disease management while awaiting study start, commercial supplies of imatinib at any dose may be prescribed to the patient but for no longer than 31 days in duration)
* Known cytopathologically confirmed Central Nervous System CNS infiltration
* Impaired cardiac function
* Severe or uncontrolled medical conditions (i.e. uncontrolled diabetes, active or uncontrolled infection)
* Acute or chronic liver, pancreatic or severe renal disease considered unrelated to disease
* Patients with another primary malignancy except if the other primary malignancy is neither currently clinically significant or requiring active intervention
* History of significant congenital or acquired bleeding disorder unrelated to cancer
* Previous radiotherapy to ≥25% of the bone marrow
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection, or gastric bypass surgery)
* Use of therapeutic coumarin derivatives (i.e. warfarin, acenocoumarol, phenprocoumon)
* Patients actively receiving therapy with strong Cytochrome P450 3A4 isoenzyme (CYP3A4) inhibitors (e.g, erythromycin, ketoconazole, itraconazole, voriconazole, clarithromycin, telithromycin, ritonavir, mibefradil)
* Patients actively receiving therapy with medications that have the potential to prolong the QT interval and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2011-01-25 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- Turkey (Türkiye) (12):
  - Novartis Investigative Site, Eskişehir, Meselik
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Bursa
  - Novartis Investigative Site, Diyarbakır
  - Novartis Investigative Site, Gaziantep
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Okmeydanı
  - Novartis Investigative Site, Talas / Kayseri
  - Novartis Investigative Site, Trabzon

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Saydam G, Haznedaroglu IC, Kaynar L, Yavuz AS, Ali R, Guvenc B, Akay OM, Baslar Z, Ozbek U, Sonmez M, Aydin D, Pehlivan M, Undar B, Dagdas S, Ayyildiz O, Akin G, Dag IM, Ilhan O. Frontline nilotinib treatment in Turkish patients with Philadelphia chromosome-positive chronic Myeloid Leukemia in chronic phase: updated results with 2 years of follow-up. Hematology. 2018 Dec;23(10):771-777. doi: 10.1080/10245332.2018.1498167. Epub 2018 Jul 11. PMID 29996726
- [Derived] Saydam G, Haznedaroglu IC, Kaynar L, Yavuz AS, Ali R, Guvenc B, Akay OM, Baslar Z, Ozbek U, Sonmez M, Aydin D, Pehlivan M, Undar B, Dagdas S, Ayyildiz O, Akkaynak DZ, Akin G, Ilhan O. Outcomes with frontline nilotinib treatment in Turkish patients with newly diagnosed Philadelphia chromosome-positive chronic myeloid leukemia in chronic phase. Hematology. 2018 Feb 27:1-7. doi: 10.1080/10245332.2018.1444919. Online ahead of print. PMID 29486663 (Retraction: PMID 29578377 Hematology. 2018 Oct;23(9):720)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 112 participants were enrolled into the study from the 15 sites in Turkey.
Pre-assignment Details: This was an open-label study with one treatment arm. The study did not involve a reference treatment.
Period: Overall Study
Arm/Group | Nilotinib
Started (participants enrolled) | 112
Completed | 92
Not Completed | 20
Not completed — Lost to Follow-up | 1
Not completed — patient not compliant with the protocol | 1
Not completed — Pregnancy | 1
Not completed — Death | 2
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 8
Not completed — progression of disease | 3
Not completed — hospitalization | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nilotinib
Number analyzed (Participants) | 112
Age, Continuous [Median (Full Range); unit: years] | 47 [19 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 63
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Major Molecular Response (MMR) During the First 12 Months
Description: Major Molecular Response (MMR) was defined as BCR-ABL1^IS ≤0.1%, on the International Scale [BCR-ABL1IS]) by 12 months. BCR is the Breakpoint Cluster Region gene / BCR gene product and ABL is the Abelson proto-oncogene. BCR-ABL is the Fusion gene from BCR and ABL/Protein product from BCR-ABL. Participants who withdrew prematurely or those who failed to provide data for the study for other reasons were designated as premature withdrawal or inevaluable, respectively, and were included in the ITT analysis as non-responders.
Time Frame: 12 months
Population: Intent-to-treat (ITT) analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 112
Participants | 74

2. Secondary Outcome: Percentage of Participants Who Achieved Major Molecular Response (MMR) up to 24 Months
Description: as for outcome 1
Time Frame: 3, 6, 9, 15, 18, 21 and 24 months
Population: ITT analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 112
Participants
  3 months | 28
  6 months | 57
  9 months | 67
  15 months | 84
  18 months | 92
  21 months | 93
  24 months | 93

3. Secondary Outcome: Percentage of Participants With Complete Cytogenetic Response (CCyR) at Month 6 and 12
Description: CCyR rate is identified as the rate of patients who had 0% of Ph+ metaphase.
Time Frame: Month 6 and 12
Population: ITT analysis set included only the participants who had measurements i.e. excluding drop outs.
Measure: Count of Participants; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 112
Participants
  Month 6: number analyzed (Participants) | 102
  Month 6 | 89
  Month 12: number analyzed (Participants) | 91
  Month 12 | 84

4. Secondary Outcome: Percentage of Participants With Complete Hematologic Response (CHR) at Month 3, 6, 9, 12, 18 and 24
Description: A confirmed complete hematological response (CHR) is defined when all of the following criteria are achieved: WBC <10 x 109/L, thrombocyte <450 x 109/L, myelocyte + metamyelocyte <%5 in blood, no sign of blast and promyelocyte in blood, basophil <%5, and no sign of extramedullary involvement.
Time Frame: Month 3, 6, 9, 12, 18 and 24
Population: ITT analysis set included only the participants who had measurements i.e. excluding drop outs.
Measure: Count of Participants; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 112
Participants
  Month 3: number analyzed (Participants) | 105
  Month 3 | 104
  Month 6: number analyzed (Participants) | 102
  Month 6 | 102
  Month 9: number analyzed (Participants) | 100
  Month 9 | 100
  Month 12: number analyzed (Participants) | 96
  Month 12 | 96
  Month 18: number analyzed (Participants) | 93
  Month 18 | 93
  Month 24: number analyzed (Participants) | 92
  Month 24 | 92

5. Secondary Outcome: Time to Major Molecular Response (MMR)
Description: Time to MMR is defined as the time period from the date of first dose intake until the first documented MMR.
Time Frame: 24 months
Population: ITT analysis set. Only participants with a MMR were included in the analysis
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Nilotinib
Number analyzed (Participants) | 93
days | 252.38 (153.22)

6. Secondary Outcome: Duration of Major Molecular Response (MMR)
Description: MMR duration is defined as the time from the date of first documented MMR to the first time of the lost MMR, progression or death.
Time Frame: 24 months
Population: ITT analysis set. Only participants with a MMR and subsequent loss of MMR were included in the analysis
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Nilotinib
Number analyzed (Participants) | 12
days | 91 (4.22)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of the treatment to end of the treatment i.e 24 months.
Arm/Group | Nilotinib
All-Cause Mortality (participants affected / at risk) | 2/112
Serious Adverse Events (participants affected / at risk) | 43/112
Other Adverse Events (participants affected / at risk) | 90/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=112)
Chest Pain (Cardiac disorders) | 3
Acute leukaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Acute myocardial infarction (Cardiac disorders) | 2
Angina unstable (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Paroxysmal arrhythmia (Cardiac disorders) | 1
Conjunctivitis allergic (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Oral disorder (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Pyrexia (General disorders) | 1
Hepatitis toxic (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Periorbital cellulitis (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Arteriogram coronary (Investigations) | 3
Lipase increased (Investigations) | 2
Weight decreased (Investigations) | 1
Lumbar vertebral fracture (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Upper limb fracture (Musculoskeletal and connective tissue disorders) | 1
Brain neoplasm (Nervous system disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin neoplasm excision (Surgical and medical procedures) | 1
Uterine dilation and curettage (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=112)
Abdominal pain upper (Gastrointestinal disorders) | 6
Alanine aminotransferase increased (Investigations) | 12
Alopecia (Skin and subcutaneous tissue disorders) | 6
Amylase increased (Investigations) | 7
Blood alkaline phosphatase increased (Investigations) | 10
Blood phosphorus decreased (Investigations) | 7
Blood triglycerides increased (Investigations) | 11
Haemoglobin decreased (Investigations) | 7
Lipase increased (Investigations) | 9
Constipation (Gastrointestinal disorders) | 7
Hyperbilirubinaemia (Hepatobiliary disorders) | 17
Hypercholesterolaemia (Hepatobiliary disorders) | 11
Influenza (Respiratory, thoracic and mediastinal disorders) | 13
Leukopenia (Blood and lymphatic system disorders) | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 16
Rash (Skin and subcutaneous tissue disorders) | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 19
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2012-05-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT01274351/Prot_000.pdf
  • Statistical Analysis Plan (2014-03-14): https://cdn.clinicaltrials.gov/large-docs/51/NCT01274351/SAP_001.pdf